CLINICAL TRIAL: NCT04181151
Title: Investigation of Activation of Latissimus Dorsi Muscle Segments During Functional Reach Activity in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuba Kaya Benli, Research Assistant, Hacettepe University
Other Study IDs: Hacettepe U
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: latissimus dorsi; stroke; electromyography; reaching activity; muscle activation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients
  Interventions: Other: Electromyographic device
- Healthy Subjects
  Interventions: Other: Electromyographic device

INTERVENTIONS:
Other: Electromyographic device — An 8-channel surface EMG system (Noraxon Telemyo DTS system, Scottsdale, USA) will be used to measure signals from muscles during surface electromyography measurements.

SUMMARY:
Latissimus Dorsi (LD); Medial sacrum, lumbar vertebrae and lower thoracic vertebrae 10-12 lateral to the spinous processus. It is a fan-like wide muscle that connects to the inferior angle of the scapula and ribs, adheres to the anterior surface of the proximal humerus and continues with aponeurosis of the contralateral Gluteus Maximus below. The activation of the LD muscle during the functional reach activity, which we use most frequently in daily living activities, affects the upper extremity and trunk movements. Therefore it is important muscle that affects the quality of movement.

The study include individuals with stroke that diagnosed by the neurologist and include healthy subjects. During sitting activity, they will be required to reach three different distances in the sagittal and scapular plane: arm length, 125% of the arm length and end point where it can reach the modified functional reach test. During the activity, electromyography (EMG) activation of latissimus dorsi, anterior deltoid and erector spina muscles will be examined with electromyographic device.

Hypothesis originating from the investigation:

H1: Latissimus dorsi muscle segments show different activation during functional reach activity.

H2: Activation of latissimus dorsi muscle segments is affected by reaching direction during functional reach activity.

H3: Activation of latissimus dorsi muscle segments is affected by reaching distance during functional reach activity.

DETAILED DESCRIPTION:
Measurements will be made during the sitting activity of the individuals included in the study. Individuals will be asked to reach midsternal height cups in two separate planes, sagittal and scapular, at arm's end, 125% of arm's distance and end point where it can reach according to modified functional reach test.

Muscle activation of latissimus dorsi, erector spina and anterior deltoid muscles will be measured by superficial electromyographic measurement. Muscle activation according to SENIAM for erector spina and anterior deltoid will be evaluated. For latissimus dorsi, activation will be measured in six segments separated according to anatomic dissection.

Reach activity will be performed 3 times on each side and at 1 minute intervals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stroke by a neurologist
* least 6 mounts after stroke
* Fugl Meyer Upper Extremity Motor Rating Scale with a value of 40 and above,
* independent sitting,
* Mini Mental Status Scale (MMSE)> 24,
* 30-67 age.

Exclusion Criteria:

* neurodegenerative disease other than stroke
* presence of neglect
* presence of apraxia
* uncorrected visual impairment
* neuromusculoskeletal pathologies
* neck and shoulder pain lasting more than 3 months

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hacettepe University Neurological Rehabilitation Unit
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Surface electromyographic measurement | 90 minutes
  Muscle activation measurement
  It is an 8-channel system for measuring signals come from muscles (Noraxon Telemyo DTS system, Scottsdale, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Tuba KAYA, R.A., Principal Investigator — Hacettepe University; Sevil BİLGİN, Assoc. Prof., Study Director — Hacettepe University; Muhammed KILINÇ, Assoc. Prof., Study Chair — Hacettepe University; Esra DÜLGER, R.A., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye/ANKARA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogduk N, Johnson G, Spalding D. The morphology and biomechanics of latissimus dorsi. Clin Biomech (Bristol). 1998 Sep;13(6):377-385. doi: 10.1016/s0268-0033(98)00102-8. PMID 11415812
- [Background] Dickstein R, Shefi S, Marcovitz E, Villa Y. Anticipatory postural adjustment in selected trunk muscles in post stroke hemiparetic patients. Arch Phys Med Rehabil. 2004 Feb;85(2):261-7. doi: 10.1016/j.apmr.2003.05.011. PMID 14966711
- [Background] Wickham JB, Brown JM. Muscles within muscles: the neuromotor control of intra-muscular segments. Eur J Appl Physiol Occup Physiol. 1998 Aug;78(3):219-25. doi: 10.1007/s004210050410. PMID 9720999
- [Background] Brown JM, Wickham JB, McAndrew DJ, Huang XF. Muscles within muscles: Coordination of 19 muscle segments within three shoulder muscles during isometric motor tasks. J Electromyogr Kinesiol. 2007 Feb;17(1):57-73. doi: 10.1016/j.jelekin.2005.10.007. Epub 2006 Feb 2. PMID 16458022
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Derived] Kaya Benli T, Kara D, Dulger E, Bilgin S. Electromyography study of six parts of the latissimus dorsi during reaching tasks while seated: A comparison between healthy subjects and stroke patients. J Electromyogr Kinesiol. 2023 Jun;70:102770. doi: 10.1016/j.jelekin.2023.102770. Epub 2023 Mar 25. PMID 37004380
- See also: SENIAM — http://seniam.org/